CLINICAL TRIAL: NCT03367000
Title: Exploring The Therapeutic Benefits Of Oral Protein Supplementation In Malnourished Dialysis Patients
Brief Title: Protein Supplementation In Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Tilakavati Karupaiah, Senior Lecturer, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF-274-2012
Record Dates: First submitted 2017-09-20; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Peritoneal Dialysis Patients
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized, open label controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceprolac (Experimental): Received supplementation which added 27.6g protein and 114kcal to daily nutritional intake as well as standard diet counselling for 6 months
  Interventions: Dietary Supplement: Ceprolac
- Dietary counseling (DC) (Placebo Comparator): Received standard diet counselling only for 6 months.
  Interventions: Other: Dietary counseling (DC)

INTERVENTIONS:
Dietary Supplement: Ceprolac — The supplement was packed into two ~15g sachets in powder form of a 90-94% whey protein isolate and hydrolysed whey. The protein powder was dissolved in 75-100ml water at room temperature and was ingested post meal once daily.
  Arms: Ceprolac
Other: Dietary counseling (DC) — Received standard dietary counseling at baseline and month 6.
  Arms: Dietary counseling (DC)

SUMMARY:
The dialysis population has a strikingly high incidence of mortality. The life expectancy of chronic dialysis patients is 20 years less than that of the general population. Approximately 50% of individuals with end stage renal disease (ESRD) die from a cardiovascular (CV) cause with mortality being 15 to 30 times higher than the age-adjusted CV mortality in the general population. There is also a steady increase of patients with diabetes and the older age groups coming into dialysis. The treatment of patients with ESRD aims at prolonging life, achieving good nutritional status and promoting the best possible functioning and quality of life (QOL). Several factors that are beyond adequacy of dialysis predict high mortality in ESRD patients. Associated co-morbidities and malnutrition factors are independently associated and the combined presence of both malnutrition and co-morbidities manifest the worst survival.Therefore this study investigates the efficacy of protein supplementation in improving health status and quality of life among peritoneal dialysis (PD) patients. This research will also generate basic data about significant health markers critical to the health status of PD patients.

DETAILED DESCRIPTION:
This study is a randomised, open labeled controlled trial where a total of 74 PD patients (37 supplemented; 37 control) were recruited from government and private settings. Subjects were randomised to either the intervention or control group. The intervention group received hydrolysed whey protein supplement and diet counselling for 6 months while the control group received only diet counselling for 6 months.

Patients who consented were first subjected to a screening for identification of eligible subjects. The screening involved basic anthropometry measures (height, weight, BMI), routine biochemistry result obtained from medical record, assessment of nutritional status and dietary evaluation. About 4ml of pre-dialysis blood was also collected by respective nurses for additional laboratory parameters (hsCRP).

During the 6 months of treatment period, patients in both control and intervention groups were assessed at baseline and end of the study (at 6 months) for anthropometry assessment, laboratory results, medical condition, hospitalisations, nutritional status, dietary intake and compliance towards supplementation (intervention group only).

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old and ≤70 years old
* Undergone dialysis at least for 6 months.
* Categorised as malnourished based on BMI <24 kg/m² and serum albumin ≤40 g/L criteria
* No incidence of hospitalisation for past 3 months, free of infection/sepsis and have not undergone surgery for past 6 months.

Exclusion Criteria:

* Patients with high inflammatory diseases, malignancy, cancer
* Vegetarian patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Serum albumin | Change from baseline serum albumin at 6 months of the study
  Biochemistry marker that indicates nutritional status
Body mass index (BMI) | Change from BMI at 6 months of the study
  Index that depicts if one's current weight is ideal for their height

CONTACTS AND LOCATIONS:
Overall Officials: Tilakavati Karupaiah, Principal Investigator — Senior Lecturer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133
- [Derived] Sahathevan S, Se CH, Ng S, Khor BH, Chinna K, Goh BL, Gafor HA, Bavanandan S, Ahmad G, Karupaiah T. Clinical efficacy and feasibility of whey protein isolates supplementation in malnourished peritoneal dialysis patients: A multicenter, parallel, open-label randomized controlled trial. Clin Nutr ESPEN. 2018 Jun;25:68-77. doi: 10.1016/j.clnesp.2018.04.002. PMID 29779821